CLINICAL TRIAL: NCT03708692
Title: The Effects of Menstrual Cycle Phases on Recovery and Cognitive Function After General Anesthesia: A Prospective, Randomized Clinical Study
Brief Title: Menstrual Cycle Phases on Recovery and Cognitive Function
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nureddin YUZKAT, Assist. Prof, Yuzuncu Yil University
Other Study IDs: Menstruel Cycle Recovery
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Menstrual Cycle; Cognitive Function; Recovery; General Anesthesia
Keywords: General Anesthesia; Recovery; Cognitive Function; Menstrual Cycle phase

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group F: Patients with menstrual cycle between 8-12 days were called Group F (Follicular phase)
  Interventions: Behavioral: Group F
- Group L: Patients with menstrual cycle between 20-24 were called Group L (Luteal phase)
  Interventions: Behavioral: Group F

INTERVENTIONS:
Behavioral: Group F — After general anesthesia, the time of return of the behaviors such as opening the eyes, fulfilling the orders or saying the age will be recorded and evaluated as the recovery criteria. In the postop recovery period, the patient will be subjected to mini mental state testing (MMST) and cognitive functions will be evaluated.
  Other Names: Group L

SUMMARY:
The aim of this study was to investigate the effects of menstrual cycle phases on recovery and cognitive function after general anesthesia.

DETAILED DESCRIPTION:
Study Protocol, Methods and Procedures to be Applied:

The study was started after obtaining the approval of the Ethics Committee, the written approvals of the patients The study is planned to conduct between October 2018- December 2018.

The study groups were selected from patients who presented to the preop anesthesia polyclinic in elective conditions, septo-rinoplasty operation under general anesthesia.

The study groups will be selected from patients who presented to the preop anesthesia polyclinic in elective conditions, septo-rinoplasty operation under general anesthesia. Assuming that there would be a 5-point difference in anxiety scores among the groups, it was decided to take 45 cases for each group with a 0.75 standard effect size, 80% power, and 5% error. Patients will be randomly assigned to 2 groups of 45 people according to their order of application. Patients will be randomized by inclusion into the determined groups. At the day of surgery, the inclusion of the patient into the one of the group will be decided.

Study inclusion criteria: The study included 80 women with ASA I-II, aged 18 to 45 years, who were accepted to participate in the study, were smoking, did not use oral contraceptives, had no menstrual irregularity (regular 28 ± 2 days menstrual cycle).

Study exclusion criteria: In preop evaluation patients had difficulties in communication, amenorrhea, pregnancy, delirium, psychological illness, major depressive disorder, patients with a history of acute illness (such as in intensive care unit follow-up), which may affect cognitive function and daily life activities in the last 6 months, malignancy, acute renal failure, substance abuse and patients older than 45 years and male sex will be excluded from the study.

Groups:

Information about menstrual cycle patterns was obtained from all cases. The days of the menstrual cycle will be determined starting from counting the first day of the last cycle. Patients with menstrual cycle between 8-12 days were called Group F (Follicular phase). Patients with menstrual cycle between 20-24 were called Group L (Luteal phase). The follow-up of the cases and the recording of the measurements were performed by an anesthesiologist who did not know which group the cases were in.

Procedures to be Applied:

Patients' gender, age, height, weight values, ASA scores, body mass index (BMI) values will be recorded.

Preoperative anesthetic examinations of the patients to be included in the study will be done at the anesthesia clinic at least 1 day before the operation. The preop tests that will be required after the examinations will consist of routine examinations.

In the operation room, hemodynamic parameters will be recorded at 5-minute intervals before induction, after intubation.

Routine procedures that is applied to similar patients will be followed during extubation of patients. The inside of the mouth will be aspirated before extubation and the patient will be extubated after muscle strength and consciousness's are restored.

Total anesthesia duration and total surgical duration, postoperative agitation, laryngospasm, hypoxia, nausea and vomiting frequency will be recorded.

After general anesthesia, the time of return of the behaviors such as opening the eyes, fulfilling the orders or saying the age will be recorded and evaluated as the recovery criteria. In the postop recovery period, the patient will be subjected to mini mental state testing (MMST) and cognitive functions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The study included 80 women with ASA I-II,
* Aged 18 to 45 years, who were accepted to participate in the study,
* were smoking,
* did not use oral contraceptives,
* had no menstrual irregularity (regular 28 ± 2 days menstrual cycle)

Exclusion Criteria:

* In preop evaluation patients had difficulties in communication,
* amenorrhea,
* pregnancy,
* delirium,
* psychological illness,
* major depressive disorder,
* patients with a history of acute illness (such as in intensive care unit follow-up),
* which may affect cognitive function and daily life activities in the last 6 months,
* malignancy,
* acute renal failure,
* substance abuse and patients older than 45 years and male sex will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study is performed on female gender with menstrual cycle.
Study Population: Current study is performed on female gender with reguler menstrual cycle, who were accepted to participate in the study,
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 1 month
  After general anesthesia, the time of return of the behaviors such as opening the eyes, fulfilling the orders or saying the age will be recorded and evaluated as the recovery criteria. In the postop recovery period, the patient will be subjected to mini mental state testing (MMST) and cognitive functions will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nureddin Yuzkat, Assist Prof, Study Chair — Yuzuncu Yil University
Locations (1):
- Van yuzuncu Yıl University, Dursun Odabas Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No